CLINICAL TRIAL: NCT07221604
Title: Setting the Agenda: An Open Pilot of a Structured Clinical Visit Agenda-Setting Intervention for Rural-Residing People With Advanced Chronic Kidney Disease
Brief Title: The Agenda-Setting for Kidney Disease Open Pilot Trial
Acronym: ASK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Catherine Hylas Saunders, Principal Scientist, Assistant Professor of Medicine and of Health Policy and Clinical Practice, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002598_2; 1K01DK139400 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease Stage 4
Keywords: Chronic kidney disease; Chronic kidney disease stage 4; Chronic kidney disease stage 5; Agenda-setting; Patient engagement; Rural; Participatory research; Open pilot
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Participation

STUDY DESIGN:
Intervention Model Description: Open feasibility pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 is Clinical Visit Agenda Setting Tool Intervention (Experimental): The study team will implement a structured clinical visit agenda-setting (SAS) intervention customized for advanced chronic kidney disease, called Chronic Kidney Disease (CKD) Topics.
  Interventions: Behavioral: Chronic Kidney Disease Structured Agenda-Setting Tool

INTERVENTIONS:
Behavioral: Chronic Kidney Disease Structured Agenda-Setting Tool — Chronic Kidney Disease (CKD) Topics is a novel clinical visit agenda-setting intervention developed through participatory research methods for people with CKD living in rural areas. CKD Topics includes 8 structured discussion topic areas with the option for patients to consider and indicate their priority topic areas and take notes before, during, and after a clinical visit.

SUMMARY:
The goal of this open pilot is to practice using an intervention and surveys before a larger pilot stepped wedge clinical trial. The intervention the researchers plan to use is Chronic Kidney Disease (CKD) Topics, and it is a structured clinical agenda-setting intervention (SAS), or a customized list of discussion topics. The people the researchers are practicing using the SAS with have advanced CKD (stages 4-5), and many of them live in rural areas. The researchers will practice administering CKD Topics, along with survey questions. By doing the open pilot, the researchers will learn if they need to modify the steps they plan to take in the larger trial.

The main questions the researchers aim to answer are:

* Do the steps for identifying eligible participants work?
* Do the steps for administering CKD Topics work?
* Do the steps to administer survey questions work?

DETAILED DESCRIPTION:
In this open pilot, the researchers will administer a novel structured agenda-setting tool (SAS) called Chronic Kidney Disease (CKD) Topics. The researchers will determine if their procedures for screening eligible participants, administering the intervention, and administering outcome and other questionnaires are appropriate. Learnings from the open pilot will feed forward into procedures in a larger planned pilot stepped wedge feasibility trial.

This study only has one arm, the intervention arm. The intervention, CKD Topics, will be administered as a quality improvement intervention.

Future Directions: This open pilot will inform procedural changes in an upcoming pilot stepped wedge feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old who have been diagnosed with advanced CKD (stages 4-5).
* Care partners, clinicians and staff supporting these CKD patients who are willing and able to provide informed consent
* English-speaking
* Able to provide informed consent
* Patient must be attending outpatient visits *(in-person and/or telehealth allowable).

Exclusion Criteria:

* Children under 18 years old will not be included
* Non-English-speaking patients and/or care partners
* Patients on dialysis
* Individuals unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Outcome: Intervention receipt | Day 1
  Our primary outcome will be feasibility, assessed by the proportion of patients who received the intervention.

OTHER OUTCOMES:
Primary Process Outcome: Enrollment Rate | Day 1
  As measured by participant enrollment in Redcap.
Preliminary Efficacy Outcome: Patient Self-Advocacy Scale (PSAS) | Day 1
  Patient Self-Advocacy Scale (PSAS); a 12-item validated scale assessing the latent construct of perceived self-advocacy for patients.
Preliminary Efficacy Outcome: Patient self-efficacy | Day 1
  Patient self-efficacy measured using the Ask, Understand, Remember Assessment, (AURA); a validated 4-item assessment of self-efficacy completed by patients.
Preliminary Efficacy Outcome: Patient self-management | Day 1
  Patient demonstration of self-management using the Perceived Medical Condition Self-Management Scale; an 8-item instrument validated to assess self-management among CKD patients; correlated with treatment adherence.
Preliminary Efficacy Outcome: Serious Illness Experience | Day 1
  Serious illness experience measured by the consideRATE questions; a validated 8-item, plain language (2nd grade) patient-reported experience measure (PREM) with Likert-like response options for patients, and care partners.
Preliminary Efficacy Outcome: Respect Experience Assessment | Day 1
  Respect experience assessment measured by the "Heard and understood" tool. Heard and Understood is a validated Single-item PREM with Likert-like response options for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
The study will use standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats, dictionaries, variable names, descriptions, and labels. An XML schema using Data Documenting Initiative standards will also be used for codebooks and other metadata as appropriate. The researchers will share RCT process and outcomes data in CSV files via openICPSR, which is a self-publishing repository for social, behavioral and health science data and part of the ICPSR.

REFERENCES:
- [Background] Brashers DE, Haas SM, Neidig JL. The patient self-advocacy scale: measuring patient involvement in health care decision-making interactions. Health Commun. 1999;11(2):97-121. doi: 10.1207/s15327027hc1102_1. PMID 16370972
- [Background] Clayman ML, Pandit AU, Bergeron AR, Cameron KA, Ross E, Wolf MS. Ask, understand, remember: a brief measure of patient communication self-efficacy within clinical encounters. J Health Commun. 2010;15 Suppl 2(Suppl 2):72-9. doi: 10.1080/10810730.2010.500349. PMID 20845194
- [Background] Frankel RM, Salyers MP, Bonfils KA, Oles SK, Matthias MS. Agenda setting in psychiatric consultations: an exploratory study. Psychiatr Rehabil J. 2013 Sep;36(3):195-201. doi: 10.1037/prj0000004. Epub 2013 Jul 1. PMID 23815174
- [Background] Gramling R, Stanek S, Ladwig S, Gajary-Coots E, Cimino J, Anderson W, Norton SA; AAHPM Research Committee Writing Group; Aslakson RA, Ast K, Elk R, Garner KK, Gramling R, Grudzen C, Kamal AH, Lamba S, LeBlanc TW, Rhodes RL, Roeland E, Schulman-Green D, Unroe KT. Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. J Pain Symptom Manage. 2016 Feb;51(2):150-4. doi: 10.1016/j.jpainsymman.2015.10.018. Epub 2015 Nov 17. PMID 26596879
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367
- [Background] Saunders CH, Durand MA, Kirkland KB, MacMartin MA, Barnato AE, Elwyn G. Psychometric assessment of the consideRATE questions, a new measure of serious illness experience, with an online simulation study. Patient Educ Couns. 2022 Jul;105(7):2581-2589. doi: 10.1016/j.pec.2022.01.002. Epub 2022 Jan 22. PMID 35260261
- [Background] Saunders CH, Durand MA, Scalia P, Kirkland KB, MacMartin MA, Barnato AE, Milne DW, Collison J, Bennett A, Wasp G, Nelson E, Elwyn G. "It helps us say what's important..." Developing Serious Illness Topics: A clinical visit agenda-setting tool. Patient Educ Couns. 2023 Aug;113:107764. doi: 10.1016/j.pec.2023.107764. Epub 2023 Apr 18. PMID 37150152
- [Background] Saunders CH, Durand MA, Scalia P, Kirkland KB, MacMartin MA, Barnato AE, Milne DW, Collison J, Jaggars A, Butt T, Wasp G, Nelson E, Elwyn G. User-Centered Design of the consideRATE Questions, a Measure of People's Experiences When They Are Seriously Ill. J Pain Symptom Manage. 2021 Mar;61(3):555-565.e5. doi: 10.1016/j.jpainsymman.2020.08.002. Epub 2020 Aug 16. PMID 32814165
- [Background] Sierpe A, Yen RW, Stevens G, Van Citters AD, Elwyn G, Saunders CH. Agenda-setting in the clinical encounter: A systematic review protocol. PLoS One. 2024 Oct 24;19(10):e0312613. doi: 10.1371/journal.pone.0312613. eCollection 2024. PMID 39446854
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Wild MG, Wallston KA, Green JA, Beach LB, Umeukeje E, Wright Nunes JA, Ikizler TA, Steed J, Cavanaugh KL. The Perceived Medical Condition Self-Management Scale can be applied to patients with chronic kidney disease. Kidney Int. 2017 Oct;92(4):972-978. doi: 10.1016/j.kint.2017.03.018. Epub 2017 May 18. PMID 28528132